CLINICAL TRIAL: NCT04886804
Title: Beamion LUNG-1: An Open Label, Phase I Dose Escalation Trial, With Dose Confirmation and Expansion, of Zongertinib (BI 1810631) as Monotherapy in Patients With Advanced or Metastatic Solid Tumors With HER2 Aberrations
Brief Title: Beamion LUNG-1: A Study to Test Different Doses of Zongertinib in People With Different Types of Advanced Cancer (Solid Tumours With Changes in the HER2 Gene)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0001; 2020-004563-47 (EudraCT Number); 2024-511246-39-00 (Registry Identifier: CTIS (EU)); U1111-1312-5969 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2021-05-04; First posted 2021-05-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neoplasm Metastasis; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase Ia - Dose escalation part (Experimental): Consecutive cohorts of patients treated with escalating doses of BI 1810631 monotherapy.
  Interventions: Drug: zongertinib
- Phase Ib - Dose expansion part: Cohort 1 (Experimental)
  Interventions: Drug: zongertinib
- Phase Ib - Dose expansion part: Cohort 2 (Experimental)
  Interventions: Drug: zongertinib
- Phase Ib - Dose expansion part: Cohort 3 (Experimental)
  Interventions: Drug: zongertinib
- Phase Ib - Dose expansion part: Cohort 4 (Experimental)
  Interventions: Drug: zongertinib
- Phase Ib - Dose expansion part: Cohort 5 (Experimental)
  Interventions: Drug: zongertinib
- Phase Ib - Dose expansion part: Cohort 6 (Experimental): Cohort only in the United States of America (USA)
  Interventions: Drug: zongertinib
- Phase Ib - Dose expansion part: Cohort 7 (Experimental): Cohort only in Japan
  Interventions: Drug: zongertinib
- Phase Ib - Dose expansion part: Cohort 8 (Experimental): Cohort only in the United States of America (USA)
  Interventions: Drug: zongertinib

INTERVENTIONS:
Drug: zongertinib — zongertinib
  Other Names: BI 1810631, Hernexeos®

SUMMARY:
The study has 2 parts. The first part is open to adults with different types of advanced cancer (solid tumours with changes in the HER2 gene) for whom previous treatment was not successful.

The second part is open to people with non-small cell lung cancer with a specific mutation in the HER2 gene.

The purpose of the first study part is to find the highest dose of a medicine called zongertinib the participants can tolerate. Once this dose is found, it will be used in the second study part to test whether zongertinib can make tumours shrink.

In this study, zongertinib is given to people for the first time. Participants take zongertinib as tablets once a day or twice a day.

The participants are in the study for as long as they benefit from and can tolerate treatment.

Study doctors regularly check the participants' health and monitor the tumours. The doctors also take note of any unwanted effects that could have been caused by zongertinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of an advanced, unresectable and/or metastatic non-haematologic malignancy. Patient must show presence of at least one measurable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
* Eastern Cooperative Oncology Group (ECOG) score of 0, 1 or 2 (ECOG=2 only for Cohorts 6 and 7) .
* Availability and patient willingness to provide a sample of tumour for confirmation of the patient´s Human epidermal growth factor receptor 2 (HER2) status. This sample can be archival material obtained at any time prior to study enrollment.
* Patient willing and able to comply with the protocol requirements for tumour biopsies (biopsies from brain metastases are not allowed).
* Adequate organ function defined as all of the following:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (≥ 1.5 x 10^3/μL) (≥ 1500/mm^3); haemoglobin ≥ 9.0 g/dL (≥ 90 g/L) (≥ 5.6 mmol/L); platelets ≥ 100 x 10^9/L (100 x 10^3/μL) (100 x 10^3/mm3) without the use of hematopoietic growth factors within 4 weeks of start of trial medication.
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), except for patients with Gilbert's syndrome: total bilirubin ≤ 3 x ULN or direct bilirubin ≤ 1.5 x ULN.
  * Estimated Glomerular Filtration Rate (eGFR) ≥ 50 mL/min - calculated using Chronic Kidney Disease Epidemiology (CKD-EPI) formula.
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN if no demonstrable liver metastases, or otherwise ≤ 5 x ULN if transaminase elevation is attributable to liver metastases.
  * Alkaline Phosphatase < 5 x ULN.
* Recovered from any previous therapy-related toxicity to ≤ Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at start of treatment (except for alopecia, stable sensory neuropathy and hypothyroidism (patients on thyroid replacement therapy) which must be ≤ CTCAE Grade 2)
* Life expectancy of at least 12 weeks at the start of treatment in the opinion of the investigator.
* At least 18 years of age at the time of consent or over the legal age of consent in countries where that is greater than 18 years.
* Signed and dated written informed consent in accordance with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Male or female patients. Women of childbearing potential (WOCBP) and men who are able to father a child must be ready and able to use highly effective methods of birth control per International Council on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.

Additional inclusion criteria for Phase Ia

* Patients with a documented diagnosis of HER2 aberration: overexpression OR gene amplification OR non-synonymous somatic mutation OR gene rearrangement involving HER2 or Neuregulin 1 (NRG1)
* Patient who has failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Patient must have exhausted, or not be a suitable candidate for, available treatment options known to prolong survival for their disease

Additional inclusion criteria for Phase Ib - Cohort 1 only

* Non-squamous non-small cell lung cancer (NSCLC) patients with documented human epidermal growth factor receptor 2 (HER2) mutation in the tyrosine kinase domain (TKD) as per local lab results.
* Patient who had received, in the advanced/metastatic setting, at least one line of systemic therapy. Patients with non-squamous NSCLC harboring additionally genomic aberrations for which approved targeted therapy is available as standard of care.

Additional inclusion criteria for Phase Ib - Cohort 2 only

* Non-squamous NSCLC patient with a documented HER2 mutation in the tyrosine kinase domain (TKD) as per local lab results.
* Treatment naïve for non-squamous NSCLC.

Additional inclusion criteria for Phase Ib - Cohort 3 only

* NSCLC Patient with a documented HER2 mutation outside of the tyrosine kinase domain (TKD) as per local lab results or squamous NSCLC patient with mutation in the TKD as per local lab results.
* Patient who had received, in the advanced/metastatic setting, at least one line of systemic therapy. Patients with NSCLC harboring additionally genomic aberrations for which approved targeted therapy is available as standard of care.

Additional inclusion criteria for Phase Ib - Cohort 4 only

* NSCLC patients with documented HER2 mutation in the TKD as per local lab results.
* NSCLC patients who are either treatment naïve or who had received any prior line of treatment, in the advanced/metastatic setting. Patients with NSCLC harboring additional genomic aberrations for which approved targeted therapy is available as standard of care.
* Patient with active brain metastases who are not eligible for immediate local therapy, as per investigator evaluation.

Additional inclusion criteria for Phase Ib - Cohort 5 only

* Non-squamous NSCLC patients with documented HER2 mutation in the TKD as per local lab results.
* Patient should have received, in the advanced/metastatic setting, at least one line of systemic therapy that includes a platinum-based combination chemotherapy and should have been treated with previous HER2 directed antibody-drug conjugates (ADC) in the same advanced/metastatic setting and developed disease progression recurrence during or after completing this therapy. Patients with NSCLC harboring additional genomic aberrations for which approved targeted therapy is available as standard of care.

Additional inclusion criteria for Phase Ib - Cohort 6 only

* Non-squamous NSCLC Patient with documented HER2 mutation in the TKD as per local lab results.
* Patient who had received, in the advanced/metastatic setting, at least one line of systemic therapy.
* Patient without active brain metastases or patient with active brain metastases who are not eligible for immediate local therapy, as per investigator evaluation.
* Patient who is not eligible for any other recruiting cohort.

Additional inclusion criteria for Phase Ib - Cohort 7 only

* Non-squamous NSCLC patient with documented HER2 mutation in the TKD as per local lab results.
* Patient who had received, in the advanced/metastatic setting, at least one line of systemic therapy.
* Patient without active brain metastases or patient with active brain metastases who are not eligible for immediate local therapy, as per investigator evaluation.
* Patient who is not eligible for any other recruiting cohort.

Additional inclusion criteria for Phase Ib - Cohort 8 only

* Treatment naïve for NSCLC
* NSCLC (adenocarcinoma or squamous) patient with documented HER2 mutation in the tyrosine kinase domain (TKD) or non-squamous NSCLC with a documented HER2 mutation in the non tyrosine kinase domain (non TKD) as per local lab results

Further inclusion criteria apply.

Exclusion Criteria:

* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to first trial treatment or planned within 6 months after screening
* Previous or concomitant malignancies other than the one treated in this trial within the last 2 years, except:

  * effectively treated non-melanoma skin cancers
  * effectively treated carcinoma in situ of the cervix
  * effectively treated ductal carcinoma in situ
  * other effectively treated malignancy that is considered cured by local treatment.
* Treatment with a systemic anti-cancer therapy or investigational drug within 21 days or 5 half-lives (whichever is shorter) of the first treatment with the study medication
* Patients who must or wish to continue the intake of restricted medication or any drug considered likely to interfere with the safe conduct of the trial
* Previous treatment with zongertinib.
* Radiotherapy within 2 weeks prior to first study treatment, except palliative radiotherapy to regions other than the chest, which is allowed up to 1 week prior to first study treatment.

Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Maximum Tolerated Dose (MTD) | At the end of Cycle 1 (each cycle is 21 days).
  Maximum tolerated dose is defined as the highest dose with less than 25% risk of the true Dose Limiting Toxicity (DLT) rate being equal to or above 33% during the MTD evaluation period in any studied regimen.
Phase Ia: Number of patients with Dose Limiting Toxicities (DLTs) in the MTD evaluation period | At the end of Cycle 1 (each cycle is 21 days).
Phase Ib - Cohorts 1, 2 and 5 : Objective response (OR) as assessed by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
  OR is defined as best overall response of complete response (CR) or partial response (PR), where best overall response is determined according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1, from the first treatment administration until the earliest of disease progression, death or last evaluable tumor assessment before start of subsequent anticancer therapy, loss to follow-up or withdrawal of consent.
Phase Ib - Cohorts 3, 6, 7, and 8: Objective response according to RECIST 1.1 by investigator assessment | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib: Cohort 4: Objective response according to Response Assessment in Neuro-Oncology for Brain Metastases (RANO-BM) by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.

SECONDARY OUTCOMES:
Phase Ia: Number of patients experiencing DLTs during the entire treatment period | From the start of the trial treatment until end of month 8, up to 8 months.
Phase Ia: Maximum measured concentration of zongertinib in plasma (Cmax) | On day 1 and on day 15 of Cycle 1 (each cycle is 21 days).
Phase Ia: Area under the concentration-time curve of zongertinib in plasma (AUC0-t2) | On day 1 and on day 15 of Cycle 1 (each cycle is 21 days).
Phase Ib - Cohorts 1, 2 and 5: Duration of objective response (DoR) according to RECIST 1.1 | From the start of the trial treatment until end of month 12, up to 12 months.
  DoR is defined as the time from first documented complete response (CR) or partial response (PR) until the earliest of disease progression or death among patients with objective response as assessed by central independent review.
Phase Ib - Cohorts 1, 2 and 5: Disease control (DC) | From the start of the trial treatment until end of month 12, up to 12 months.
  DC is defined as best overall response of complete response (CR) or partial response (PR) or stable disease (SD) where best overall response is defined according to RECIST version 1.1 as assessed central independent review, from first treatment administration until the earliest of disease progression, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up or withdrawal of consent.
Phase Ib - Cohorts 1, 2 and 5: Progression-free survival (PFS) | From the start of the trial treatment until end of month 12, up to 12 months.
  PFS is defined as the time from first treatment administration until tumor progression according to RECIST version 1.1 as assessed by central independent review, or death from any cause, whichever occurs earlier.
Phase Ib - Cohorts 1, 2 and 5: Objective response according to response assessment in neuro-oncology for brain metastases (RANO-BM) criteria as assessed by central independent review for patients with central nervous system (CNS) lesions at baseline | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohorts 1, 2 and 5: Disease control according to RANO-BM criteria as assessed by central independent review for patients with CNS lesions at baseline | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohorts 1, 2 and 5: Objective response according to RECIST 1.1 criteria as assessed by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohorts 1, 2 and 5: Disease control according to RECIST 1.1 criteria as assessed by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohorts 3, 6, 7 and 8: Duration of objective response according to RECIST 1.1 by investigator assessment | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohorts 3, 6, 7 and 8: Disease control according to RECIST 1.1 as assessed by the investigator | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohorts 3, 6, 7 and 8: Progression-free survival according to RECIST 1.1 as assessed by the investigator | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohorts 3, 6, 7 and 8: Objective response according to RANO-BM criteria as assessed by the investigator for patients with CNS lesions at baseline | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohorts 3, 6, 7 and 8: Disease control according to RANO-BM criteria as assessed by the investigator for patients with CNS lesions at baseline | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: Duration of objective response (DoR) according to RANO-BM by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: Disease control (DC) according to RANO-BM by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: Progression-free survival (PFS) according to RANO-BM as assessed by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: DoR according to RECIST 1.1 by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: DC according to RECIST 1.1 by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: PFS according to RECIST 1.1 as assessed by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: OR according to RECIST 1.1 by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: Duration of OR according to RECIST 1.1 by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - Cohort 4: PFS according to RECIST 1.1 by central independent review | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - All cohorts: Overall survival (OS), defined as time from first treatment administration until death from any cause | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - All Cohorts: Number of patients experiencing DLTs during the entire treatment period | From the start of the trial treatment until end of month 12, up to 12 months.
Phase Ib - All Cohorts: Change from baseline to Day 1 of Cycle 5 in EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) physical functioning domain score | Baseline and on Day 1 of Cycle 5 (each cycle is 21 days).
Phase Ib - All Cohorts: Change from baseline to Day 1 of Cycle 5 in Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) total score | Baseline and on Day 1 of Cycle 5 (each cycle is 21 days).
Phase Ib - All Cohorts: Change from baseline to Day 1 of Cycle 5 in EORTC item List 46 (IL46) score | Baseline and on Day 1 of Cycle 5 (each cycle is 21 days).

CONTACTS AND LOCATIONS:
Locations (85):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Precision NextGen Oncology, Beverly Hills, California
  - City of Hope-Duarte-56419, Duarte, California
  - City of Hope - Seacliff, Huntington Beach, California
  - City of Hope-Irvine-69674, Irvine, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California Irvine, Orange, California
  - University of California Davis, Sacramento, California
  - Georgetown University, Washington D.C., District of Columbia
  - Holy Cross Hospital-Fort Lauderdale-57892, Fort Lauderdale, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Hawaii Cancer Care - Honolulu, Honolulu, Hawaii
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Sarah Cannon Research Institute-Nashville-48456, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Macquarie University, Macquarie Park, New South Wales, Australia
- Ordensklinikum Linz GmbH, Linz, Austria
- Brussels - HOSP Jules Bordet, Anderlecht/Brussels-Capital, Belgium
- China (15):
  - Beijing Cancer Hospital, Beijing
  - Jilin Province Cancer Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - Fujian Cancer Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The Affiliated Cancer Hospital, Guangxi Medical University, Nanning
  - Shanghai Chest Hospital, Shanghai
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital Affiliated Tongji Medical College Huazhong University of S & T, Wuhan
  - First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- France (6):
  - HOP Louis Pradel, Bron
  - CTR Leon Berard, Lyon
  - HOP Timone, Marseille
  - INS Curie, Paris
  - HOP Pontchaillou, Rennes
  - INS Gustave Roussy, Villejuif
- Germany (5):
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Köln (AöR), Cologne
  - Technische Universität Dresden, Dresden
  - Justus-Liebig Universität Gießen, Giessen
  - Pius-Hospital, Oldenburg, Oldenburg
- Hong Kong (2):
  - Prince of Wales Hospital-Hong Kong-20715, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Israel (4):
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center Tel HaShomer, Tel Litwinsky
- Italy (3):
  - Istituto Di Candiolo, Candiolo (TO)
  - Istituto Nazionale IRCCS Tumori Fondazione Pascale, Napoli
  - Azienda Ospedaliera Unversitaria di Parma, Parma
- Japan (7):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Shikoku Cancer Center, Ehime, Matsuyama
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osaka, Sakai
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - National Cancer Center Hospital, Tokyo, Chuo-ku
- Netherlands (2):
  - Nederlands Kanker Instituut, Amsterdam
  - Leids Universitair Medisch Centrum (LUMC), Leiden
- Hospital CUF Porto, Porto, Portugal
- Singapore (2):
  - National University Hospital-Singapore-22806, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (5):
  - Chungbuk National University Hospital, Chungju
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario De Valencia, Valencia
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden
- United Kingdom (3):
  - The Royal Marsden Hospital, Chelsea, London
  - Hammersmith Hospital, London
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Heymach JV, Ruiter G, Ahn MJ, Girard N, Smit EF, Planchard D, Wu YL, Cho BC, Yamamoto N, Sabari JK, Zhao Y, Tu HY, Yoh K, Nadal E, Sadrolhefazi B, Rohrbacher M, von Wangenheim U, Eigenbrod-Giese S, Zugazagoitia J; Beamion LUNG-1 Investigators. Zongertinib in Previously Treated HER2-Mutant Non-Small-Cell Lung Cancer. N Engl J Med. 2025 Jun 19;392(23):2321-2333. doi: 10.1056/NEJMoa2503704. Epub 2025 Apr 28. PMID 40293180
- [Derived] Heymach JV, Opdam F, Barve M, Tu HY, Wu YL, Berz D, Schroter L, Botilde Y, Sadrolhefazi B, Serra J, Yoh K, Yamamoto N. HER2-Selective Tyrosine Kinase Inhibitor, Zongertinib (BI 1810631), in Patients With Advanced/Metastatic Solid Tumors With HER2 Alterations: A Phase Ia Dose-Escalation Study. J Clin Oncol. 2025 Apr 10;43(11):1337-1347. doi: 10.1200/JCO-24-01727. Epub 2025 Mar 3. PMID 40030100
- [Derived] Heymach J, Opdam F, Barve M, Gibson N, Sadrolhefazi B, Serra J, Yamamoto N. A Phase I, Open-Label, Dose Confirmation, Escalation, and Expansion Trial of BI 1810631 as Monotherapy in Patients With Advanced or Metastatic Solid Tumors With HER2 Aberrations. Clin Lung Cancer. 2023 Mar;24(2):e65-e68. doi: 10.1016/j.cllc.2022.10.008. Epub 2022 Nov 11. PMID 36528522
- See also: Related Info — http://www.mystudywindow.com